CLINICAL TRIAL: NCT04292548
Title: Salivary TAS, TOS, LL-37 and Dental Status in Passive Smoking Children
Status: Completed | Type: Observational
Sponsor: Merve Erkmen Almaz (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Sponsor-Investigator, Merve Erkmen Almaz, Assist prof, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: Kırıkkale pediatric dentistry
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Passive Smoking; Oxidative Stress; Dental Caries; Children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group (passive smoking children)
  Interventions: Diagnostic Test: taking saliva samples to determine TAS, TOS and LL-37
- control group
  Interventions: Diagnostic Test: taking saliva samples to determine TAS, TOS and LL-37

INTERVENTIONS:
Diagnostic Test: taking saliva samples to determine TAS, TOS and LL-37

SUMMARY:
The aim of the present study was to determine the effect of passive smoking on the levels of salivary TAS, TOS, LL-37 and dental status in children.In the study the parents of children were asked to fill out a complete survey about smoking habits. After filling out the questionnaire, according to the survey results, a total of 180 children were included to the study as follows; 90 children exposed to passive smoking, and 90 children in the control group (unexposed controls). Also demographic data were recorded (age, gender, parental education levels, child's tooth-brushing habit and child's daily dietary sugar exposure, family income). Dental examination of children were performed and caries prevalance of the patients were recorded. Unstimulated saliva samples were collected from children. Saliva 'cotinine levels' which are expected to increase in passive smoking group; 'antimicrobial peptide LL-37' and oxidative stress markers 'total antioxidant status' (TAS), and' total oxidant status' (TOS) were evaluated by using Enzyme-linked immunosorbent assay (ELISA). The obtained data parameters of the two groups were evaluated and comparison was performed.

ELIGIBILITY:
Inclusion Criteria:

-Systemically healthy children

Exclusion Criteria:

* The presence of orthodontic / intraoral appliance
* Any disease or condition known to affect defense system
* Uncooperative children

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children, referring for dental examination to the Department of Pediatric Dentistry of Kirikkale University, were selected.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
salivary oxidative stress values: TAS level | 1 day (once after the dental examination)
  Unstimulated saliva samples were collected from children.
salivary oxidative stress values: TOS level | 1 day (once after the dental examination)
  Unstimulated saliva samples were collected from children.
salivary LL-37 level | 1 day (once after the dental examination)
  Unstimulated saliva samples were collected from children.
salivary cotinine levels | 1 day (once after the dental examination)
  Unstimulated saliva samples were collected from children for describing passive smoking children.

IPD SHARING:
Plan to Share IPD: No
As soon as possible data will be shared when it is published in a journal.